CLINICAL TRIAL: NCT05028153
Title: Azithromycin Treatment of Hospitalized Children With Asthmatic Symptoms: A Double-blinded, Randomized, Controlled Study
Brief Title: Azithromycin Treatment of Hospitalized Children With Asthmatic Symptoms
Acronym: COPSACazt
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Copenhagen Studies on Asthma in Childhood (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-20065249
Record Dates: First submitted 2021-08-19; First posted 2021-08-31 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Childhood Asthma With Acute Exacerbation
Keywords: Asthma; Infections; Wheeze; Antibiotics
MeSH Terms: conditions — Asthma; Infections; Respiratory Sounds

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antibiotics (Active Comparator): Azithromycin (10mg/kg) administered via oral suspension for 3 consecutive days
  Interventions: Drug: Azithromycin Oral Liquid Product
- Placebo (Placebo Comparator): Placebo with no active substance administered via oral suspension for 3 consecutive days
  Interventions: Other: Placebo mixture

INTERVENTIONS:
Drug: Azithromycin Oral Liquid Product — 10 mg/kg for 3 consecutive days
  Arms: Antibiotics
Other: Placebo mixture — Placebo mixture containing no active substance
  Arms: Placebo

SUMMARY:
The purpose of this double-blind, randomized, controlled clinical trial is to investigate the effect of a three-day azithromycin treatment versus placebo treatment in children aged 1-5 years who are hospitalized due to asthma-like symptoms.

DETAILED DESCRIPTION:
The children who are included must be have a known history with one or more previous episodes of asthmatic symptoms and is currently / have received treatment with SABA as monotherapy or SABA in combination with ICS and possibly LTRA. The primary purpose during hospitalization is to replicate the results of our previous study, where it was shown that azithromycin treatment significantly shortened the duration of the asthmatic episode. In this study, hospitalized children who provide a more diverse group than the COPSAC2010 cohort will be included. In addition, the study aims to focus on examining the individual response to treatment. The expectation is that in the future the study will be able to contribute to personal treatment based on the child's respiratory microbiome and / or immunological profile so that only the children who will benefit from the azithromycin treatment will receive it. The expectation is also that the study will contribute to an increased understanding of the influence of bacteria on asthma-like episodes in preschool children, and thus will lead to an evidence-based better treatment of these.

The study hypothesis is:

● that antibiotic treatment with azithromycin compared to placebo in the patient group aged 1-5 years, known with previous episode (s) with asthma-like symptoms and is currently / have received treatment with SABA as monotherapy, or SABA in combination with ICS and possibly LTRA, will lead to a significant reduction in the symptom burden and duration of the asthmatic episode in days.

ELIGIBILITY:
Inclusion Criteria:

* Previous episode(s) with asthma-like symptoms and / medical treatment with SABA as mono-therapy or SABA in combination with ICS and possibly LTRA.
* The parent/guardian(s) agrees to admit the child and is willing to follow the procedure of the trial.
* The child is between 12-71 months old.
* Fluent Danish skills with parents / guardians.

Exclusion Criteria:

* Known allergy to macrolide antibiotics.
* Known impaired liver function.
* Known renal impairment.
* Known with neurological or psychiatric diseases.
* Known with congenital or documented acquired QT interval.
* Known for clinically relevant bradycardia, cardiac arrhythmia or severe heart failure.
* Clinical signs of pneumonia (Objective findings, including severe tachypnoea: respiratory rate (RF)> 50 and / or Fever: temperature> 39 °C and / or C-reactive protein (CRP)> 50).

Ages: 12 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2022-11-14 (Actual); Primary Completion 2026-11-13 (Estimated); Study Completion 2032-11-13 (Estimated)

PRIMARY OUTCOMES:
Duration in days of the asthma-like episode from the start of randomization. | 1-30 days
  Number of days based on a diary.

SECONDARY OUTCOMES:
Change in symptom score. | From day 1 after randomization to completion of each randomized asthmatic episode aged 1-5 years.
  Using a previously validated symptom scoring model based on a diary. The score range is from 0 (no symptoms) and up to 3 (depending on presence of one or more of the followings symptoms: Cough, breathlessness and wheezing).
Effect modification in relation to the child's respiratory microbiota profile. | Sample time, day 1
  Airway microbiota, pathogenic bacteria and vira as measured by 16S-rRNA and whole genome sequencing.
Effect modification in relation to the child's respiratory immunological profile. | Sample time, day 1
  Evaluation of immune mediator profiles (cytokine and chemokine levels) in the upper airway epithelial lining fluid.
The length of hospitalization (days) | 1-30 days
  Determined by participants medical record.
Need for SABA during the asthma-like episode | 1-30 days
  Number of days based on a diary.
Need for oral corticosteroids (OCS) during the asthma-like episode. | 1-30 days
  Number of days based on a diary.
Stratification of the above analyzes. | Sample time, day 1
  On the basis of the presence or absence of bacteria/microbiota in the respiratory tract, based on outcomes 3, 4 and 5.
Number of days away from daycare offers. | 1-30 days
  Number of days based on a diary.
Health economic gain based on treatment costs and lost earnings. lost earnings for parent / guardian (s) | 1-30 days
  The number of days home from daycare causing parent absenteeism due to illness based on this diary registration.
Gut microbiome profile | 1-30 days
  Occurrence, diversity and abundance of gut microbiota using 16S rRNA sequencing and whole genome sequencing.
Resistance profiles | 1-30 days
  Occurrence, diversity and abundance of antibiotic resistance genes as assessed by metagenome sequencing.
Adverse Event (AE) registration | 1-30 days
  Number of events and type of event based on a diary.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Stokholm, MD, PhD, Principal Investigator — University Hospital of Copenhagen, DK-2820 Gentofte, Denmark
Locations (1):
- University Hospital of Copenhagen, Gentofte Municipality, Denmark

REFERENCES:
- [Derived] Kyvsgaard JN, Ralfkiaer U, Folsgaard N, Jensen TM, Hesselberg LM, Schoos AM, Bonnelykke K, Bisgaard H, Stokholm J, Chawes B. Azithromycin and high-dose vitamin D for treatment and prevention of asthma-like episodes in hospitalised preschool children: study protocol for a combined double-blind randomised controlled trial. BMJ Open. 2022 Apr 13;12(4):e054762. doi: 10.1136/bmjopen-2021-054762. PMID 35418427